CLINICAL TRIAL: NCT05919004
Title: Uncontrolled Postviral Asthma in Patients With Long Covid
Brief Title: Uncontrolled Postviral Asthma and Persistent Symptoms After COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: The Norwegian Sports Medicine Centre - Football Association, Oslo, Norway (Other)
Responsible Party: Principal Investigator, Tonje Reier-Nilsen, MD PhD, The Norwegian Sports Medicine Centre - Football Association, Oslo, Norway
Other Study IDs: IdrettensHelsesenter
Record Dates: First submitted 2023-06-22; First posted 2023-06-26 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Long COVID
Keywords: postviral asthma; diagnosis; long covid; telemedicine; lung function; digital spirometer
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: App-based spirometer — App-based spirometer to perform serial spirometry to assess lung function variatione

SUMMARY:
Patients with long covid referred for physical rehabilitation at the Norwegian Sports Medicine Centre - Football Association in Oslo, Norway, were assessed for postviral asthma.

DETAILED DESCRIPTION:
All patients performed methacholin bronchial provocation test, and those with a negative bronchial provocation were eqipped with an app-based spirometer to detect excessive lung variability. Eventual detection of postviral asthma will be treated according to GINA guidelines and eventual effect will be assessed by lung function variability and symptoms.

ELIGIBILITY:
Inclusion Criteria:

° Patients with long covid for more than 6 months referred for physical rehabilitation

Exclusion Criteria:

° None

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with long covid for more than 6 months
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Excessive lung function variation | 8 months
  Lung function given as FEV1.
Perceived symptoms of long covid | 8 months
  On a Likert scale 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Idrettens Helsesenter, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No